CLINICAL TRIAL: NCT01998334
Title: Continuous Blood Purification for Regulation of Early Inflammatory Response In Severe Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP BUNDLE-CRRT; 12411950500 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2013-11-10; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Acute Pancreatitis
Keywords: Systemic Inflammatory Response Syndrome; Continuous Blood Purification
MeSH Terms: conditions — Pancreatitis; Systemic Inflammatory Response Syndrome | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CVVH 6h (Experimental): CVVH 6h for first three days
  Interventions: Other: CVVH 6h
- CVVH 10h (Experimental): CVVH 10h for first three days
  Interventions: Other: CVVH 10h
- CVVHDF (Experimental): CVVHDF 6h for first three days
  Interventions: Other: CVVHDF 6h

INTERVENTIONS:
Other: CVVH 6h — CVVH 6h for first three days
  Arms: CVVH 6h
Other: CVVH 10h — CVVH 10h for first three days
  Arms: CVVH 10h
Other: CVVHDF 6h — CVVHDF 6h for first three days
  Arms: CVVHDF

SUMMARY:
Systemic Inflammatory response syndrome(SIRS) is common in patients with severe acute pancreatitis (SAP) in early stage. Continuous Blood Purification (CBP), especially Continuous Veno-Venous Hemofiltration(CVVH) is proved to have an important role in SAP patients to control SIRS. But the detail treatment for this is controversial. In this study, the investigators aim to evaluate the different effects of three kinds of treatment protocols which is CVVH 6h,continuous venovenous hemodiafiltration(CVVHDF) 6h,CVVH 10h for first three days in SAP patients. Compare the vital sign, SIRS parameters, and others between these three groups. This study will try to find a better way for CBP in patients with SAP

DETAILED DESCRIPTION:
Condition Severe Acute Pancreatitis

Intervention CVVH 6 hours for first three days CVVH 10 hours for first three days CVVHDF 6 hours for first three days

All therapeutic volume is 45ml/kg.h, Device: Braxter HF 1200

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Diagnosis of pancreatitis:

   * Typical pain
   * Increase in serum lipase or amylase
   * Onset of abdominal pain within <=72h before admission
2. The diagnosis criteria of Severe Acute Pancreatitis is according to Atlanta criteria revisited in 2012
3. no chronic diseases such as Chronic Obstructive Pulmonary Disease, Diabetes Mellitus and so on
4. Age from 18 to 65 years old

Besides criteria above, the patient should also satisfied one of these CBP criteria:

1. Have Acute Kidney Injury satisfied RIFLE classification (risk above): increased Serum Creatinine > 1.5 times baseline，26.5umol/L increase, or urine output < 0.5ml/kg.h for 6 hours
2. Systemic Inflammatory Response Syndrome: temperature >38℃ or<36℃；heart rate respiratory rate White blood cell count >12*10^9/L，or< 4*10^9/L
3. Refractory acid-base and electrocyte balance disorder, metabolic acidosis conservative treatment is not effective.

Exclusion Criteria:

1. Pregnancy
2. Chronic pancreatitis
3. Immunosuppression condition such as HIV, Corticosteroid for 3 weeks in 60 days; White Blood Cell < 0.5*10^9/L for 10 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The Efficiency of CBP with Inflammatory Response | 3 days
  Efficiency of CBP with inflammatory response was assessed by the following measurements:
  1. Inflammatory mediators removal:tumor necrosis factor-α, interleukin(IL-1, IL-2, IL-6, and IL-8, IL-10, sIL-2R)before and after CBP in first three days
  2. SIRS parameters variation: (Heart rate, respiratory rate, White Blood Cell, Temperature, C response protein) before and after CBP in first three days

SECONDARY OUTCOMES:
mortality | 28 days
  Mortality of 28 days
operation time | 28 days
  operation time of 28 days
local complication of severe acute pancreatitis | 28 days
  local complication of SAP in 28 days

OTHER OUTCOMES:
ICU and hospital duration | participants will be followed for the duration of hospital stay, an expected average of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enqiang Mao, M.D, Study Director — Department of EICU Ruijin Hospital
Locations (1):
- Department of EICU, Ruijin Hospital,, Shanghai, Shanghai Municipality, China